CLINICAL TRIAL: NCT02578459
Title: A Pilot Study to Evaluate the Efficacy of ITDD vs. CMM in the Treatment of Pancreatic Cancer Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never initiated by sponsor. Patients where never recruited.
Sponsor: Flowonix Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM-02
Record Dates: First submitted 2015-10-14; First posted 2015-10-19 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2018-07

CONDITIONS: Pain Management; Cancer Pain
Keywords: Cancer pain; Intrathecal therapy; Pain; Pancreatic cancer
MeSH Terms: conditions — Agnosia; Cancer Pain; Pain; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intrathecal Drug Delivery (ITDD) (Experimental): These subjects will have a Prometra System implanted and managed with the appropriate drug regimen to treat their pain.
  Interventions: Device: Intrathecal Drug Delivery System
- Conventional Medical Management (CMM) (Active Comparator): These subjects will be treated with conventional medical management to treat their pain.
  Interventions: Other: Conventional Medical Management

INTERVENTIONS:
Device: Intrathecal Drug Delivery System — The Prometra Pump is a battery-operated, implantable, programmable infusion pump that dispenses pain medication into the intrathecal space through an implanted infusion catheter.
  Other Names: Prometra Programmable Infusion System
  Arms: Intrathecal Drug Delivery (ITDD)
Other: Conventional Medical Management — Treatment with conventional medical management will include using standard systemic pain medications such as narcotics, nonsteroidal anti-inflammatory drugs (NSAIDs), and neuropathic medications (examples: gabapentin, Lyrica, Cymbalta) that are typically used to treat pancreatic cancer pain.
  Arms: Conventional Medical Management (CMM)

SUMMARY:
The purpose of this study is to compare efficacy of pain treatment with ITDD to efficacy of pain treatment with CMM in patients with pancreatic cancer pain.

DETAILED DESCRIPTION:
This study is a non-randomized, open-label, single-center study that will compare efficacy of pain treatment with ITDD to efficacy of pain treatment with CMM in patients suffering from pancreatic cancer pain.

There will be two treatment groups: Study group (ITDD): These subjects will have a Prometra System implanted and managed with the appropriate drug regimen to treat their pain. Systemic analgesics will not be prescribed for this group. Control group (CMM): These subjects will be treated with CMM to treat their pain.

A maximum of 30 subjects (maximum of 15 in each treatment group) may be enrolled in this study at one study center.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has Stage IV pancreatic cancer.
2. Patient agrees not to be treated by other oncologists or anesthesiologists during the study.
3. Patient agrees not to obtain pain medications from other physicians during the study.
4. Patient is at least 22 years of age.
5. Investigator considers the patient to be able and willing to fulfill all study requirements.
6. Patient is able to understand the study and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Patient meets any of the contraindications for use of the Prometra Programmable Infusion System (for patients in the ITDD group).
2. Patient is enrolled in another clinical study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale Pain Scores | Three months
  Level of pain is rated on the visual analog scale. Pain scores after three months of therapy will be compared to baseline pain scores to see if there is a difference.

SECONDARY OUTCOMES:
Survival Rates | Two years
  Data will be analyzed to test for correlation between survival and pain scores, and survival rates and treatment type.
Quality of Life Scores | Two years
  Difference in quality of life between treatment groups.
Cancer Treatments | Two years
  Difference between treatment group in the number of cancer treatment initiated during the study
Hospitalizations and Emergency Room Visits | Two years
  Difference between treatment group in the number of times they are hospitalized or visit the emergency room during the study
Adverse Events | Two years
  Adverse events reported by each treatment group will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Kloster, MD, Principal Investigator — Menorah Medical Center
Locations (1):
- Menorah Medical Center, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Dr. Daniel R. Kloster — https://menorahmedicalcenter.secure.ehc.com/physicians/profile/Daniel-R-Kloster-MD
- See also: Dr. Jaswinder Singh — https://researchmedicalcenter.secure.ehc.com/physicians/profile/Jaswinder-Singh-MD